CLINICAL TRIAL: NCT00256971
Title: Functioning Balance in Patients After Surgery for Torn Meniscus: Meniscectomy vs Meniscal Repair; A Prospective Study
Brief Title: Balance in Patients After Surgery for Torn Meniscus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: MEN-BM-HMO-CTIL
Record Dates: First submitted 2005-11-20; First posted 2005-11-22 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2005-11

CONDITIONS: Torn Menisci
MeSH Terms: interventions — Meniscectomy

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: meniscectomy

SUMMARY:
The important role of the menisci in knee function and in preserving knee health has been shown in several studies. Additionally to principal functions of load transmission and shock absorption, meniscus contributes to knee joint proprioception and probably also to joint stability.Study about affect of meniscus injury on balance posture has not previously been published.Surgical practice is increasingly aimed at minimal resection of injured tissue, preserving a stable meniscal remnant with as much function as possible.The purpose of this study is to determine whether menisci surgery have any effects on relatively new postural control measures, in correlation with functional balance assessment. The second purpose is to establish the affect of different types of menisci surgery on balance impairment (meniscectomy vs tear repair), in correlation with a long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Participants have to be healthy people
* 18-40 years old
* After a traumatic event of only one knee

Exclusion Criteria:

* Previous knee surgery
* OA per arthroscopy
* Neurological problem
* Any other orthopedic problem of lower limbs
* Systemic arthritic condition (RA, SLE etc.)
* Severe cognitive problem with restricted consent
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-11; Study Completion 2008-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: isabella schwartz, Principal Investigator — Hadassah Medical Organization IRB
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel